CLINICAL TRIAL: NCT05140785
Title: In Vivo Molecular Mapping of Adult Primary Brain Tumour Activity Using Novel Magnetic Resonance Imaging (MRI): a Pilot Study
Brief Title: Mapping Molecular Markers of Brain Tumour Activity Using MRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Erasmus Medical Center (Other); King's College London (Other)
Responsible Party: Principal Investigator, Thomas Booth, Chief Investigator and Consultant Diagnostic and Interventional Neuroradiologist, Department of Neuroradiology, Ruskin Wing, King's College Hospital NHS Foundation Trust, London. SE5 9RS, King's College Hospital NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 288219
Record Dates: First submitted 2021-11-10; First posted 2021-12-01 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain tumour patients (Experimental): Patients will be those undergoing routine care of primary brain tumours. Study group patients will undergo additional MRI sequences and biopsies in addition to the standard of care.
  Interventions: Diagnostic Test: Advanced MRI sequences

INTERVENTIONS:
Diagnostic Test: Advanced MRI sequences — Advanced MRI sequences which look to a) determine structure of a primary brain tumour and b) metabolism within a primary brain tumour

SUMMARY:
Regions of tumour whose cells (the building blocks of the tumour) are actively multiplying generate a particular type of molecular footprint (consisting of various types of proteins) compared to tumours whose cells are relatively stable. In addition, tumour cells begin to develop a network of blood vessels that not only supply them with nutrients and oxygen, but also provide a pathway for tumour spread. There is a critical period between when these proteins and blood vessel network develops, and when tumour growth is visible using current MRI scanning. Therefore, making the process of tumour activity visible on clinical MRI scans is an important step in demonstrating and anticipating tumour growth. The study aims to do this by utilising various novel and non-invasive MRI techniques.

This project is a collaboration between research groups at King's College London (UK) and the Erasmus University Rotterdam (The Netherlands). The novel MRI techniques will be incorporated into the pre-surgical imaging protocol of patients with primary brain tumours. The images will be compared with molecular measurements made from biopsies taken during surgery to show that they accurately map where activity is high and low within the tumour.

DETAILED DESCRIPTION:
Patients recruited into this study will be those for whom a surgical resection or biopsy of a primary brain tumour has already been planned by the King's College Hospital Neuro-oncology team. All patients in the UK arm of this international study will be recruited at the King's College Hospital site. Research imaging performed on patients enrolled in this study will take place at the Guy's and St Thomas' Hospital site.

For patients who have consented to be included in our research study, novel MRI techniques will be included in addition to the standard primary brain tumour imaging protocol, to provide additional information about the nature of the primary tumour: for example, the structural components and metabolism.

The MRI scan will last approximately 60 minutes, which is approximately 30 minutes longer than the standard brain tumour biopsy protocol. Further MRI scans will be performed after surgery and, if necessary, at recurrence (up to a maximum of three scans per patient) to look at advanced imaging changes at each time-point alongside structural changes. These additional scans should also last a maximum of 60 minutes.

All patients will undergo surgery for biopsy/resection of the tumour as part of the standard of care. All routine surgical procedures, pre-surgical and post-surgical care will take place predominantly at King's College Hospital site. Before craniotomy takes place for tumour resection, the neurosurgeon will take 3 tissue samples of the tumour. This will occur via stereotactic (computer-guided) biopsies. A needle will be guided through to a location of interest determined by the novel MRI techniques. This should result in an extension of the surgery time of approximately 30 minutes (10 minutes per biopsy), in addition to the approximately 4 hours needed for the surgery.

After removal, each biopsy specimen is put into a suitable container for preservation. The container will be de-identified and shipped to the Department of Pathology, Erasmus University Rotterdam, The Netherlands where the specimen will be securely stored.

The samples will be cut and slide-mounted for staining. When looking at the specimen under a microscope, particular features which suggest how aggressive the tumour is will be looked for. Information gathered from the tissue biopsies will then be compared and matched to information on the original MRI scan to see whether the novel images obtained can accurately predict the aggressiveness of different parts of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of 18 years or older
* Referred for surgery (resection or biopsy) of primary brain tumour
* Written informed consent

Exclusion Criteria:

* Contra-indication for MRI contrast
* Inability to give consent
* Have received/are receiving chemotherapy at time of MRI
* Patient is pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of the MRI signal intensity (advanced MRI sequence 1; arbitrary units) and glioma protein concentration (g/L) in a 1 x 1 x 1 cm region of interest (R value) | 5 years
  MRI signal will be recorded from different regions of interest within a glioma where stereotactic surgical biopsies taken and protein concentration determined.

SECONDARY OUTCOMES:
Correlation of the MRI signal intensity (advanced MRI sequence 2; arbitrary units) and glioma metabolite concentration (g/L) in a 1 x 1 x 1 cm (R value) | 5 years
  MRI signal will be recorded from different regions of interest within a glioma where stereotactic surgical biopsies taken and metabolite concentration determined.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Booth, PhD, Principal Investigator — King's College London
Locations (1):
- King's R&I department, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No